CLINICAL TRIAL: NCT06262477
Title: A Randomized, Double-Blind, Parallel-Group, Phase I Study to Evaluate the Pharmacokinetics, Safety and Immunogenicity of BIIB800 s.c. Compared to Actemra® in Healthy Male Participants
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Immunogenicity of BIIB800 Subcutaneously (SC) Compared to Actemra® in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL-TCZ-12280
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB800 (Experimental): Participants will receive a single dose of BIIB800 via autoinjector, administered SC in the outer area of the upper arm on Day 1 of the study.
  Interventions: Drug: BIIB800
- Actemra (Experimental): Participants will receive a single dose of Actemra via autoinjector, administered SC in the outer area of the upper arm on Day 1 of the study.
  Interventions: Drug: Actemra

INTERVENTIONS:
Drug: BIIB800 — Administered as specified in the treatment arm.
  Other Names: BAT1806
  Arms: BIIB800
Drug: Actemra — Administered as specified in the treatment arm.
  Other Names: Tocilizumab; RoActemra
  Arms: Actemra

SUMMARY:
The primary objective of the study is to show equivalence in pharmacokinetics (PK) of BIIB800 and Actemra following SC administration of a single dose to healthy male participants. The secondary objective of the study is to evaluate PK over time, clinical safety, pharmacodynamic (PD) profiles and immunogenicity of BIIB800 and Actemra.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index between 18.5 and 29.9 kilograms per meter square (kg/m^2), inclusive.
* Total body weight between 60.0 and 90.0 kg, inclusive.
* Systolic blood pressure <135 millimeters of mercury (mmHg) or >85 mmHg at Screening, after being supine for at least 5 minutes.
* No clinically significant (as determined by the Investigator) 12-lead electrocardiogram (ECG) abnormalities, no cardiac pacemaker.

Key Exclusion Criteria:

* History or positive test result at Screening for human immunodeficiency virus (HIV).
* History of hepatitis C infection or positive test result at Screening for hepatitis C virus antibody.
* Current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and total hepatitis B core antibody [anti-HBc]).
* Serious infection (as determined by the Investigator) within the 6 months prior to Screening.
* History of systemic hypersensitivity reaction to the active drug substance, the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study.
* History of immunodeficiency or other clinically significant immunological disorders, or autoimmune disorders.
* History of clinically significant (in the opinion of the Investigator) atopic allergy (e.g., asthma, urticaria, eczematous dermatitis, allergic rhinitis), hypersensitivity, or allergic reactions.
* History of angioedema.
* A positive diagnostic tuberculosis test result within 35 days prior to Day -1, defined as a positive QuantiFERON® test result or 2 successive indeterminate QuantiFERON test results.
* Any prior exposure to tocilizumab or to any other agent directly acting on IL-6 or on its receptors including investigational products (e.g., siltuximab, sarilumab etc.).
* Administration of immunoglobulins for anti-tetanus and anti-rabies post-exposure prophylaxis within 3 weeks prior to administration of study drug.
* Any live or attenuated immunization or vaccination given within 30 days prior to Day -1 or planned to be given during the study period.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (3):
  - Fortrea Clinical Research Unit Inc., Daytona Beach, Florida
  - Fortrea Clinical Research Unit Inc., Dallas, Texas
  - Fortrea Clinical Research Unit Inc., Madison, Wisconsin
- Fortrea Clinical Research Unit Inc., Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male participants were enrolled in this study from 02 January 2024 to 04 October 2024 at investigative sites in the US and UK.
Pre-assignment Details: Overall, 342 participants were screened, of which 300 were randomized in the study. Of the 300 participants randomized, 150 participants received a single dose of BIIB800 subcutaneous (SC) injection and 150 participants received a single dose of Actemra SC injection.
Groups:
- BIIB800: Participants received a single dose of BIIB800 via autoinjector, administered SC in the outer area of the upper arm on Day 1 of the study.
- Actemra: Participants received a single dose of Actemra via autoinjector, administered SC in the outer area of the upper arm on Day 1 of the study.
Period: Overall Study
Arm/Group | BIIB800 | Actemra
Started | 150 | 150
Completed | 149 | 148
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The all participants analysis set (APAS) included all participants who provided informed consent and had any protocol-led assessment recorded in the study clinical database (i.e., excluded screen failures).
Groups:
- Total: Total of all reporting groups
Arm/Group | BIIB800 | Actemra | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (9.34) | 34.0 (9.93) | 33.9 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 150 | 150 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 39
  Not Hispanic or Latino | 130 | 130 | 260
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 108 | 108 | 216
  Race: Black or African American | 23 | 25 | 48
  Race: Asian | 10 | 11 | 21
  Race: Multiple | 8 | 5 | 13
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Tocilizumab
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: The pharmacokinetic analysis set (PKAS) included all randomized study participants with at least one evaluable pharmacokinetic (PK) parameter. 'Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliter (μg/mL)
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 148
micrograms per milliter (μg/mL) | 10.5 (43.3) | 10.0 (41.3)
Statistical Analysis 1: Comparison: BIIB800 vs Actemra; Test type: Equivalence — The natural log (ln)- transformed Cmax was analysed using analysis of covariance (ANCOVA) model, which included actual treatment & body weight category (<75 kilograms [kg], ≥75 kg) as factors. The ratio of geometric least square means (GLSM), and corresponding confidence interval (CI) was obtained by taking the exponential of the differences in LSMs and corresponding CIs on the ln scale; Ratio of GLSM = 1.05, 90.3% CI 2-sided [0.974 to 1.13]

2. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tocilizumab
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: The PKAS included all randomized study participants with at least one evaluable PK parameter. 'Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)*μg/ mL
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 133 | 137
hours (h)*μg/ mL | 2380 (44.9) | 2240 (41.1)
Statistical Analysis 1: Comparison: BIIB800 vs Actemra; Test type: Equivalence — The natural log (ln)- transformed AUC0-inf was analyzed using ANCOVA model, which included actual treatment & body weight category (<75 kg, ≥75 kg) as factors. The ratio of GLSM, and corresponding CI was obtained by taking the exponential of the differences in LSMs and corresponding CIs on the ln scale; Ratio of GLSM = 1.07, 90.3% CI 2-sided [0.988 to 1.15]

3. Primary Outcome: Area Under the Concentration-Time Curve up to the Last Measurable Concentration (AUC0-t) of Tocilizumab
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/ mL
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 148
h*μg/ mL | 2120 (45.9) | 2000 (44.0)
Statistical Analysis 1: Comparison: BIIB800 vs Actemra; Test type: Equivalence — The natural log (ln)- transformed AUC0-t was analyzed using ANCOVA model, which included actual treatment & body weight category (<75 kg, ≥75 kg) as factors. The ratio of GLSM, and corresponding CI was obtained by taking the exponential of the differences in LSMs and corresponding CIs on the ln scale; Ratio of GLSM = 1.06, 90.3% CI 2-sided [0.985 to 1.15]

4. Secondary Outcome: Time to Reach Cmax (Tmax) of BIIB800 and Tocilizumab
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 148
hours | 84.0 [12.1 to 241] | 96.0 [24.0 to 168]

5. Secondary Outcome: Apparent Total Body Clearance (CL/F) of BIIB800 and Actemra
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 133 | 137
Liter per hour (L/h) | 0.0680 (44.9) | 0.0723 (41.1)

6. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of BIIB800 and Actemra
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 133 | 137
hours | 68.5 [36.3 to 202] | 68.3 [33.0 to 151]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious AEs (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant who has received a pharmaceutical product, regardless of causal relationship with the product. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease which is temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE was defined as an AE that starts during or after dosing or starts prior to dosing and increases in severity after dosing. An SAE is any untoward medical occurrence that results in death, in the view of the Investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, is a medically important event.
Time Frame: From the first dose of study drug up to the end of the study (up to Day 57)
Population: The safety analysis set (SAFS) included all randomized study participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 150
Participants
  TEAEs | 76 | 86
  TESAEs | 2 | 0

8. Secondary Outcome: Area Under the Effect-Time Curve (AUE) of Soluble Interleukin-6-Receptor (sIL-6R)
Description: sIL-6R levels were determined using a validated immunoassay method based on ProteinSimple Ella.
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: The pharmacodynamics analysis set (PDAS) included all randomized study participants with at least one evaluable pharmacodynamic (PD) parameter i.e., sIL-6R and/or high sensitivity C-reactive protein (hsCRP). 'Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 149
hours*nanograms per milliliter (h*ng/mL) | 209000 (68400) | 202000 (58200)

9. Secondary Outcome: Maximum Observed Effect (Emax) of sIL-6R
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: The PDAS included all randomized study participants with at least one evaluable PD parameter i.e., sIL-6R and/or hsCRP. 'Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 149
ng/mL | 459 (99.1) | 452 (90.6)

10. Secondary Outcome: Time to Emax (tEmax) of sIL-6R
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 149
hours | 336 [4.00 to 1370] | 336 [144 to 1350]

11. Secondary Outcome: AUE of High Sensitivity C-Reactive Protein (hsCRP)
Description: hsCRP was determined using a particle enhanced immunoturbidometric assay.
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours*milligrams per liter (h*mg/L)
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 142 | 140
hours*milligrams per liter (h*mg/L) | 1190 (1480) | 1780 (2570)

12. Secondary Outcome: Minimum Observed Effect (Emin) of hsCRP
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 142 | 140
milligrams per liter (mg/L) | 0.133 (0.124) | 0.131 (0.105)

13. Secondary Outcome: Time to Emin (tEmin) of hsCRP
Time Frame: Pre-dose on Day 1 and multiple time points post-dose (up to Day 57)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 142 | 140
hours | 72.0 [0 to 483] | 96.0 [0 to 338]

14. Secondary Outcome: Number of Participants With Positive Tocilizumab Anti-drug Antibodies (ADA) and Neutralizing Antibodies (nAb) Status
Description: The ADA-positive status was determined as a participant with either a pre-existing ADA-positive status (an ADA-positive sample at baseline [prior to administration of study treatment]) or a treatment-induced ADA-positive status (a participant with a negative ADA sample at baseline [pre-dose] and at least one ADA-positive sample after the administration of the study treatment. The nAb-positive status was determined in the same manner that of ADA status. ADA and nAb were analyzed in human serum using validated electrochemiluminescence (ECL) assays based on the MesoScale Discovery platform and were measured using validated ECL methods.
Time Frame: Day 1 to Day 57
Population: The SAFS included all randomized study participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 150 | 150
Participants
  ADA | 26 | 12
  nAb | 21 | 9

15. Secondary Outcome: Geometric Mean Titer of Anti-drug Antibodies (ADA)
Description: ADA titre was defined as a quasi-quantitative expression of the level of ADA in a sample.
Time Frame: Pre-dose, Days 15, 29, 57
Population: The SAFS included all randomized study participants who received the study drug. 'Overall number of participants analyzed' indicates the number of participants with positive ADA. 'Number analyzed (n)' signifies the number of participants evaluable for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titre
Arm/Group | BIIB800 | Actemra
Number analyzed (Participants) | 26 | 12
titre
  Pre-dose: number analyzed (Participants) | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 3
  Day 15 |  | 160.0 (0.0)
  Day 29: number analyzed (Participants) | 3 | 3
  Day 29 | 201.6 (41.7) | 254.0 (94.7)
  Day 57: number analyzed (Participants) | 26 | 10
  Day 57 | 477.3 (96.7) | 452.5 (152.4)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to the end of the study (up to Day 57)
Description: The SAFS included all randomized study participants who received the study drug. Treatment-emergent adverse events are reported.
Arm/Group | BIIB800 | Actemra
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 2/150 | 0/150
Other Adverse Events (participants affected / at risk) | 75/150 | 86/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB800 (N=150) | Actemra (N=150)
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB800 (N=150) | Actemra (N=150)
Headache (Nervous system disorders) | 13 | 16
Dizziness (Nervous system disorders) | 3 | 4
Lethargy (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2
Brain fog (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Piriformis syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 8
Injection site bruising (General disorders) | 6 | 5
Influenza like illness (General disorders) | 1 | 4
Pyrexia (General disorders) | 2 | 1
Injection site pain (General disorders) | 2 | 1
Vessel puncture site bruise (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site swelling (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 4 | 3
Rhinitis (Infections and infestations) | 5 | 2
Nasopharyngitis (Infections and infestations) | 1 | 5
Pharyngitis (Infections and infestations) | 0 | 2
Balanitis candida (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Norovirus infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 25
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 3 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 7
Neutrophil count decreased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT06262477/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT06262477/SAP_001.pdf